CLINICAL TRIAL: NCT04746274
Title: The More the Merrier and Brevity is the Soul of Wit? Efficacy of a Multicomponent Positive Psychological Intervention Conducted in an Online Large-group One-session Format
Brief Title: An Online Large-group One-session Training to Enhance Positive Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Svenja Schaumburg, Research Fellow / PhD Student, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 683
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Psychology, Positive; Psychological Distress
Keywords: large-group intervention; one-session intervention; positive mental health; positive psychological intervention; positive psychology; wellbeing; online intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online large-group one-session multicomponent positive psychological intervention (Experimental)
  Interventions: Behavioral: Online large-group one-session multicomponent positive psychological intervention
- Online large-group one-session cognitive intervention targeting dysfunctional thoughts (Active Comparator)
  Interventions: Behavioral: Online large-group one-session cognitive intervention targeting dysfunctional thoughts
- Waitlist Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Online large-group one-session multicomponent positive psychological intervention — The intervention is aimed at enhancing positive mental health by using components from positive psychology or positive psychotherapy. These include for exapmle using character strengths, savoring the moment, goal setting and goal attainment. The intervention is conducted in an online group format via videoconference with a duration of approximately 3 and a half hours.
  Arms: Online large-group one-session multicomponent positive psychological intervention
Behavioral: Online large-group one-session cognitive intervention targeting dysfunctional thoughts — The intervention is aimed at reducing dysfunctional thoughts by applying strategies known from the cognitive therapy of depression. These include for example identification of automatic thoughts and cognitive biases as well as evaluating evidence for and against automatic thoughts. The intervention is conducted in an online group format via videoconference with a duration of approximately 3 and a half hours.
  Arms: Online large-group one-session cognitive intervention targeting dysfunctional thoughts

SUMMARY:
Current models suggest that mental health is not the mere absence of a mental disorder. Rather, mental health consists of two factors, mental disorder symptoms and positive mental health, that can be regarded as continua. Programmes applying interventions known from the positive psychology or positive psychotherapy framework have been shown to enhance psychological wellbeing, subjective wellbeing and to reduce depressive symptoms. However, interventions were mostly conducted in an individual or small group setting and usually consisted of more than one session. The few trainings of minimal length that were conducted in group settings only used one intervention strategy or one part of multicomponent positive psychological interventions. Therefore, the conclusions that can be drawn regarding the effectiveness of short group-interventions are limited. In this study, the investigators plan to conduct an online large-group one-session training to enhance positive mental health that comprises multiple positive psychological interventions (e.g. character strengths, positive communication, goal attainment, etc). Furthermore, an active as well as a passive (waitlist) control group are included in the study. In the active control group, dysfunctional thoughts are adressed that are known to everybody but exist in a great measure in people suffering from depressive disorders. Methods used in cognitive therapy are applied in this group. Participants will be recruited from a community sample without any inclusion criteria but being of legal age. The only exclusion criterion is not having the appropriate technical equipment for participation in a videoconference. Positive mental health as well as other constructs of mental health will be assessed before and after training and at one month and six months follow up to investigate long-term effects of the intervention.

DETAILED DESCRIPTION:
In general, the investigators expect an increase in positive mental health in the multicomponent positive psychological intervention (MPPI) group. This effect should be present at the assessment points one month and six months after training. Furthermore, the increase in positive mental health in the MPPI group is expected to be larger than in the two control groups (cognitive intervention targeting dysfunctional thoughts [CIDT], waitlist). Furthermore, the investigators hypothesize participants to benefit from the MPPI in terms of other constructs related to mental health, i.e. self efficacy, happiness, wellbeing, positive emotions, and life satisfaction, in the long term. This increase is expected to be larger in the MPPI than in the two control groups. A decrease in depressive symptoms is hypothesized to occur in the MPPI as well as in the CIDT group.

The sample under investigation will be a community sample. All participants can attain the training for free and there is no payment for participation. One week before the first training day, the random allocation to the three groups will take place. Two days before the first training day, all participants are asked to fill out another survey through a link sent to them via e-mail. This survey comprises all outcome measures. The same procedure is carried out one day after, one month after and six months after the first training day. After the last assessment time point, the training for the waitlist control group will be conducted.

The target sample size is 300 participants (100 per group). The investigators will attempt to recruit more participants, assuming that not all will complete the study, especially the assessment after six months.

The investigators used the software program G*Power to conduct a power analysis. The goal was to obtain .95 power to detect a small effect size of .1 at the standard .05 alpha error probability. The investigators extended the calculated sample size of 264 participants to a target sample size of 300 participants as there was no study before that compared an online multicomponent large-group one-session training to enhance positive mental health with an online large-group one-session intervention targeting dysfunctional thoughts. Therefore, the effect size for the comparison of these two groups could be smaller than f = .1.

The primary outcome measure will be analyzed with a 3x2 repeated measures ANOVA.

For all other outcome measures, the investigators will use 3 x 4 between-within repeated measures ANOVAs (rmANOVA) to analyze the results. The first factor is a between-subjects factor that comprises the three groups MPPI, CIDT and waitlist control group. The second factor is a within-subjects factor reflecting the four assessment time points two days before the intervention, one day after the intervention, one month after the intervention and six months after the intervention. This analysis will be conducted for positive mental health, life satisfaction, affect, generalized self-efficacy, happiness, wellbeing, stress perception, positive and negative aspects of mental health, depression, anxiety and stress, social support and media-related variables. Before these analyses are carried out, correlations among the outcome measures are calculated. If outcome measures correlate significantly high (above .5), they will be first analyzed together in a between-within repeated measures MANOVA to control for alpha-error accumulation. After that, the separate analyses will be conducted. Furthermore, there will be paired comparisons between each of the three groups, reducing the first between-subjects factor in the between-within rm(M)ANOVA to two levels. For each group, rmANOVAs will be conducted to analyze the change of outcome variables over time entailing paired contrasts between the assessment time points.

ELIGIBILITY:
Inclusion Criteria:

• Aged 18 years or above

Exclusion Criteria:

• Not having the appropriate technical equipment for participation in a videoconference

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-10-17 (Actual)

PRIMARY OUTCOMES:
change on positive mental health scale (german version; Lukat, Margraf, Lutz, van der Feld, & Becker, 2015) | two days before the intervention and one month after the intervention
  9 items, 4-point Likert scale, large change in a positive direction means better outcome

SECONDARY OUTCOMES:
change on positive mental health scale (german version; Lukat, Margraf, Lutz, van der Feld, & Becker, 2015) | two days before the intervention, one day after the intervention, one month after the intervention (already specified as primary outcome measure), six months after the intervention
  9 items, 4-point Likert scale, large change in a positive direction means better outcome
change on generalized self efficacy scale (german version; Schwarzer & Jerusalem, 1999) | two days before the intervention, one day after the intervention, one month after the intervention, six months after the intervention
  10 items, 4-point Likert scale, large change in a positive direction means better outcome
change on satisfaction with life scale (german version; Glaesmer, Grande, Braehler, & Roth, 2011) | two days before the intervention, one day after the intervention, one month after the intervention, six months after the intervention
  5 items, 7-point Likert scale, large change in a positive direction means better outcome
change on subjective happiness scale (Lyubomirsky & Lepper, 1999; german version) | two days before the intervention, one day after the intervention, one month after the intervention, six months after the intervention
  4 items, 7-point Likert scale, large change in a positive direction means better outcome
change on positive and negative affect schedule (german version; Breyer & Bluemke, 2016) | two days before the intervention, one day after the intervention, one month after the intervention, six months after the intervention
  20 items, 5-point Likert scale, two subscales negative affect: large change in a negative direction means better outcome positive affect: large change in a positive direction means better outcome
change in the degree of subjectively experienced stress concerning a specific situation measured with the questionnaire "primary appraisal secondary appraisal" (PASA; german version; Gaab, 2009) | two days before the intervention, one day after the intervention, one month after the intervention, six months after the intervention
  The questionnaire assesses the two processes proposed in Lazarus' transactional model of stress: primary appraisal and secondary appraisal. Each process is operationalized by two subscales (yielding four level 1 subscales and two level 2 subscales). The subscales will be analyzed seperately and a stressindex will be calculated by calculating the difference between primary and secondary appraisal.
  16 items, 6-point Likert-scale, for the stressindex, large changes in a negative direction mean better outcome
change on mental health continuum - short form (Keyes et al., 2008; german translation) | two days before the intervention, one day after the intervention, one month after the intervention, six months after the intervention
  14 items, 6-point Likert scale, three subscales emotional wellbeing, subjective wellbeing and personal wellbeing, large change in a positive direction means better outcome
change on general health questionnaire (german version; Linden et al., 1996) | two days before the intervention, one day after the intervention, one month after the intervention, six months after the intervention
  12 items, 4-point Likert scale, large change in a negative direction means better outcome
change on depression anxiety stress scale (DASS-21; german version; Nilges & Essau, 2015) | two days before the intervention, one day after the intervention, one month after the intervention, six months after the intervention
  21 items, 4-point Likert scale, 3 subscales that are analyzed separately (depression, anxiety, stress), large change in a negative direction means better outcome
change on brief form of the perceived social support questionnaire (german version; Lin, Hirschfeld, & Margraf, 2019) | two days before the intervention, one day after the intervention, one month after the intervention, six months after the intervention
  6 items, 5-point Likert scale, large change in a positive direction means better outcome
change of frequency of media use (TV, internet, gaming, smartphone, social media) | two days before the intervention, one day after the intervention, one month after the intervention, six months after the intervention
  7-point scale for each medium, large change in a negative direction means better outcome
change of use of social media (frequency of social media use of different platforms, e.g. facebook, tumblr; accesses per day; time per day) | two days before the intervention, one day after the intervention, one month after the intervention, six months after the intervention
  frequency: 7-point scale, accesses per day and time per day measured continously, large change in a negative direction means better outcome
change on brief version of the Bergen Social Media Addiction Scale (german version; Brailovskaia, Schillack, & Margraf, 2020) | two days before the intervention, one day after the intervention, one month after the intervention, six months after the intervention
  6 items, 5-point Likert scale, large change in a negative direction means better outcome

OTHER OUTCOMES:
general rating of success | one day after the intervention
  how helpful was the training for you (0 = not helpful at all; 10 = extremely helpful); how successful was the training for you ( 0 = not successful at all; 10 = extremely successful); did the training meet your expectations (0 = did not meet my expectations at all; 10 = met all my expectations); would you recommend the training to a friend (0 = would not recommend it; 10 = would absolutely recommend it)
practice / use of the learned strategies | one month after the intervention, six months after the intervention
  how often did you practice / use the learned strategies (0 = never; 10 = always)
helpfulness of the learned strategies | one month after the intervention, six months after the intervention
  how helpful was the use of the learned strategies (0 = not helpful at all; 10 = extremely helpful)

CONTACTS AND LOCATIONS:
Overall Officials: Svenja Schaumburg, M. Sc., Principal Investigator — Ruhr University of Bochum
Locations (1):
- Ruhr-University of Bochum, Bochum, Germany

IPD SHARING:
Plan to Share IPD: Yes
It is planned to make individual participant data available on publication of the associated study results, via a publically-available data repository such as Open Science Framework. Data made available will be the research data reported in the publication, with the exception of any data that could compromise participant anonymity.